CLINICAL TRIAL: NCT05143320
Title: Cognitive and Neuropsychiatric Features of COVID-19 Patients After Hospital Dismission: an Italian Sample.
Brief Title: Cognitive, Emotional and Behavioural Impairments in Patients After Sars-Cov2 Infection
Status: Completed | Type: Observational
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Other Study IDs: NPS impairment in Covid-19
Record Dates: First submitted 2021-12-02; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: COVID-19; Sars-CoV-2 Infection
Keywords: Covid-19; Cognition; Teleneuropsychology; Memory; Executive Functions
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid+
- Covid-

SUMMARY:
Recent studies suggest cognitive, emotional and behavioural impairments occur in patients after SARS-CoV-2 infection. Problems with memory, attention, information processing and executive functions are particularly prevalent in these patients, probably due to hypothesised sensitivity of the hippocampus to the virus. Cognitive impairment is also present in patients with no neurological, neuropsychological and neuropsychiatric history. Therefore, the aim of the present study is to describe neuropsychological and neuropsychiatric features in patients recovered from moderate to severe forms of Covid-19 some weeks after hospital dismission.

ELIGIBILITY:
Inclusion Criteria:

* Positive PCR from nasopharyngeal swab
* No ICU admission

Exclusion Criteria:

* Diagnosis of neurologic or psychiatric disorders;
* Previous cognitive impairment;
* Other medical conditions negatively affecting the cognitive status.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who were hospitalized in the Covid ward and recovered from the acute phase of Covid-19 with no need of ICU admission. All patients had SARS-Cov-2 infection confirmed by positive PCR from nasopharyngeal swab. Neuropsychological study was performed on average 20 days after hospital discharge to have the most recent possible cognitive profile related to the infection. We enrolled 29 healthy controls (Covid-) who did not have SARS COV 2 infections with a 1:1 match by age, education and gender.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Cognitive and neuropsychiatirc symptoms in Covid-19 patients | About 20 days after hospital dismission
  Prevalence of neuropsychological and neuropsychiatric impairment in patients after hospitalization in patients with Sars-Cov2 infection.

CONTACTS AND LOCATIONS:
Locations (1):
- "Moriggia Pelascini" Hospital, Gravedona, Como, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cian V, De Laurenzis A, Siri C, Gusmeroli A, Canesi M. Cognitive and Neuropsychiatric Features of COVID-19 Patients After Hospital Dismission: An Italian Sample. Front Psychol. 2022 May 24;13:908363. doi: 10.3389/fpsyg.2022.908363. eCollection 2022. PMID 35686079